CLINICAL TRIAL: NCT05543330
Title: A Phase 1, Multicenter, Open-label, Dose-increasing Study to Evaluate the Safety, Tolerability, PK/PD and Preliminary Efficacy of M701, a Recombinant Epcam and CD3 Bispecific Antibody , in Patients With Malignant Pleural Effusions Caused by NSCLC
Brief Title: A Phase Ib/II Clinical Trial of M701 in the Treatment of Malignant Pleural Effusions Caused by NSCLC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wuhan YZY Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M70103
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Malignant Pleural Effusions; NSCLC Stage IV
Keywords: Malignant Pleural Effusions; NSCLC
MeSH Terms: conditions — Pleural Effusion, Malignant; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: For Phase 2 study, the patients are enrolled into 2 arm parallelly.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Pleural drainage and M701 infusion
  Interventions: Drug: M701 pleural infusion; Procedure: Pleural drainage
- Control group (Sham Comparator): Pleural drainage only or plus chemotherapy as investigator's choice.
  Interventions: Procedure: Pleural drainage; Drug: Cisplatin pleural infusion

INTERVENTIONS:
Drug: M701 pleural infusion — M701 pleural infusion on Days 1,4,7 and 10.
  Arms: Experimental group
Procedure: Pleural drainage — Pleural effusion drainage via Ultra-sound guidance on Day 1.
Drug: Cisplatin pleural infusion — Cisplatin pleural infusion (30-50mg/m2) on Day 1.
  Arms: Control group

SUMMARY:
This is a phase 1/phase 2, multicenter, open-label study to evaluate the safety, tolerability, PK, PD, immunogenicity and preliminary efficacy of M701 in patients with treatment of malignant pleural effusions caused by NSCLC.

DETAILED DESCRIPTION:
This study is consisted of two phase, Phase Ib and II:

Phase 1b includes dose escalation phase and cohort expansion phase. In dose escalation phase, up to 4 dose-escalation cohorts will be sequentially enrolled with regular "3+3" design. DLTs will be evaluated during the first treatment cycle, which is 28 days. In cohort expansion phase, after the RP2D was identified, participants were enrolled in an open-ended manner. Participants were assigned to groups A(3 injections), B (4 injections)and C(6 injections) on a 1:1:1 basis to evaluate the dose frequency.

Phase II:The dose and dosing frequency of M701 drug for the Phase II clinical trial were determined based on a combination of the tolerance1 and efficacy of M701 in the Phase Ib trial. Then the participants were randomly divided into two groups: the test group(M701) and the control group(cisplatin or pleural effusions suctions). The pleural effusions response (ORR) and Puncture Free Survival （PuFS）will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged > 18 years.
2. Histologically- or cytologically-confirmed non-small cell lung cancer that has progressed after first line systemic therapy.
3. Malignant pleural effusion diagnosed histologically or cytologically, with moderate or above moderate pleural fluid (sitting pleural fluid depth ≥ 4 cm via ultrasound, expected pleural fluid volume ≥ 500 mL) . Require clinical intervention and not treated yet.
4. Patients who have an washout period of ≥ 4 weeks or 5 half-life of the drug (including radiotherapy, chemotherapy, immunotherapy, biologic, targeted, hormonal therapy, and 14 days for local radiotherapy) between the last systemic therapy and the first dose; however, no washout period is required if the subject has new pleural fluid or poor control of current pleural fluid after at least 2 cycle systemic therapy.
5. Patients who had recovered to grade 0-1 of any toxic reaction to prior antineoplastic therapy as determined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) V5.0, with the exception of alopecia, hyperpigmentation and ≤ grade 2 neuropathy, hormone replacement hypothyroidism or other adverse events confirmed to have turned chronic.
6. Patients with physical status ECOG score (PS) of 0-2.
7. Patients with life expectancy ≥ 12 weeks.
8. Bone marrow: absolute neutrophil count (ANC) ≥ 1.5 ×10^9/L, platelet count ≥ 100 ×10^9/L, hemoglobin ≥ 8.5 g/dL (without blood transfusion within14 days of the first dose of study drug); Liver: bilirubin (TBIL)≤ 1.5 x upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤ 3 x ULN ( ≤ 5 x ULN in case of liver metastases); Kidney: serum creatinine ≤1.5 x ULN.
9. Patients must understand and voluntarily sign the written informed consent.

Exclusion Criteria:

1. Patients with asymptomatic pleural fluid and not requiring clinical intervention, or bilateral malignant pleural fluid, or proposed perfusion of the chest cavity presenting with pleural fluid separation.
2. Patients with central nervous system (CNS) metastases resulting in clinical symptoms or requiring therapeutic intervention; patients previously treated for brain metastases may be enrolled if they have been asymptomatic for ≥ 4 weeks prior to the first dose and have imaging indicating stable disease and do not require corticosteroid or anticonvulsant therapy.
3. Patients with a known history of severe allergy to M701 drug components or antibody-like macromolecular drugs.
4. Patients with contraindications to thoracentesis.
5. Patients who have undergone major surgical procedures within 4 weeks prior to the first dose.
6. Patients with extensive liver metastases (>70%).
7. Patients with uncontrollable active infection (NCI-CTCAE V5.0 ≥ grade 2).
8. Patients required long-term hormonal or immunosuppressive therapy, e.g. active autoimmune disease, maintenance therapy after organ transplantation, except that the following are allowed to enter screening: type I diabetes mellitus, hypothyroidism that can be controlled by replacement therapy only, skin diseases that do not require systemic therapy (e.g. vitiligo, psoriasis or alopecia).
9. Patients with severe respiratory disease which, in the judgment of the investigator, makes them unsuitable for entry; or combined interstitial pneumonia.
10. Patients with history of severe cardiovascular disease, including previous coronary artery bypass grafting or coronary stenting, myocardial infarction within 6 months, congestive heart failure (New York Classification of Cardiac Function Class III-IV) or unstable angina, or uncontrolled hypertension.
11. Patients with QTc interval > 480 ms,family or personal history of long or short QT syndrome, clinically significant history of ventricular arrhythmias or implantation of a defibrillation device for ventricular arrhythmias.
12. Patients with a history of (non-study tumour) malignancy (except squamous and basal cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or other, non-invasive lesions that the investigator and sponsor agree have been cured and have a minimal risk of recurrence within 3 years) within 3 years prior to the date of first study drug administration.
13. Patients who have active hepatitis B (HBV-DNA quantification ≥ 1 x 10^4 copies/mL or 2000 IU/mL), active hepatitis C (positive for hepatitis C antibodies and HCV-RNA above the lower limit of detection of the assay), active syphilis with positive HIV antibodies.
14. Pregnant or breastfeeding woman,Plan to conceive within six months;
15. Patients with a confirmed history of neurological or mental disorders, including epilepsy and dementia.
16. Those that are deemed ineligible for this clinical trial by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) | From the time of the first dose (Day 1) until the forth dosing (Day 28)
  Dose limiting toxicities during the first 28 days after the first administrations of study drug in each cohort.
Incidence of AEs | From the start of administration to the end of the study or 28 days after the administration is stopped
  Incidence and severity of AEs, including but not limited to vital signs, physical examination, laboratory tests. All AEs will be classified as Grades 1 through 5 as defined by NCI CTCAE v5.0.
Objective Response Rate(4 weeks/8 weeks) of pleural effusion | From the time of first dosing (Day 1) until disease progression(up to 56 days)
  the rate of patients with pleural effusion CR and PR at 4 weeks / 8 weeks, based on CT evaluation .

SECONDARY OUTCOMES:
Area under the curve (AUC) of M701 | From the time of first dosing (Day 1) until disease progression or toxicity intolerance(up to 16 days)
  The endpoints for assessment of PK of M701 include serum concentrations of M701 at different timepoints after M701 administration.
Maximum observed concentration (Cmax) of M701 | From the time of first dosing (Day 1) until disease progression or toxicity intolerance(up to 16 days)
  The endpoints for assessment of PK of M701 include serum concentrations of M701 at different timepoints after M701 administration.
Minimum observed concentration (Cmin) of M701 | From the time of first dosing (Day 1) until disease progression or toxicity intolerance(up to 16 days)
  The endpoints for assessment of PK of M701 include serum concentrations of M701 at different timepoints after M701 administration.
Half-time (t1/2) of M701 | From the time of first dosing (Day 1) until disease progression or toxicity intolerance(up to 16 days)
  Half-time (t1/2) of M701
Anti-drug antibodies(ADAs) titer | From the time of first dosing (Day 1) until disease progression or toxicity intolerance(up to 16 days)
  The immunogenicity of M701 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).
Neutralizing antibody titer | From the time of first dosing (Day 1) until disease progression or toxicity intolerance(up to 16 days)
  The immunogenicity of M701 will be collected by testing the antibody titer of the neutralizing antibody.
Concentrations of tumor biomarker in pleural effusions | From the time of first dosing (Day 1) until disease progression or toxicity intolerance(up to 56 days)
  As tumor biomarkers, concentrations of CEA, CyFra21-1, SCC and NSE in malignant pleural effusions will be examined at Day 1 and Day10.
Expression level of EpCAM-positive cells in pleural effusions | From the time of first dosing (Day 1) until disease progression (up to 56 days)
  The number and expression levels of EpCAM-positive cells in pleural effusions will be measured by pathological methods (including cytospin, immunohistochemical techniques, etc.)
Ratio of EpCAM-positive tumour cell/leucocyte | From the time of first dosing (Day 1) until disease progression (up to 56 days)
  Ratio of EpCAM positive tumour cell/leucocyte in pleural effusions will be measured by FACS method.
Rate of with successful pleurodesis (4/8 weeks) | From the time of first dosing (Day 1) until disease progression (up to 56 days)
  the rate of patients with successful pleurodesis at 4 weeks / 8 weeks
Puncture-free survival rate at 4/8 weeks | From the time of first dosing (Day 1) until disease progression (up to 56 days)
  the rate of patients without extra puncture at 4/8 weeks after the initial drainage.
Pleural signs and symptoms | From the time of first dosing (Day 1) until disease progression (up to 56 days)
  Using the Lister Quadruple Scale to record pleural effusions at 4 weeks/ 8 weeks.

OTHER OUTCOMES:
Objective Response Rate of Tumor | From the time of first dosing (Day 1) until disease progression (up to 56 days)
  ORR is defined as percentage of participants who achieved complete response (CR), partial response (PR), based on RESIST 1.1 .
Disease Control Rate of tumor | From the time of first dosing (Day 1) until disease progression (up to 56 days)
  ORR is defined as percentage of participants who achieved complete response (CR), partial response (PR), and stable disease (SD), based on RESIST 1.1 .
Duration of disease control(DDC) | 12 months (anticipated)
  Duration of disease control(DDC) was calculated from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, based on RESIST 1.1 .
Progression-free disease survival (PFS) | 12 months (anticipated)
  PFS was defined as the time between the date of first dose of M701 and either disease progression or death, whichever occurs first.
Half-year / One-year Survival Rates | 12 months (anticipated)
  Survival Rates at 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yiping Zhang, Principal Investigator — Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital); Zhengbo Song, Principal Investigator — Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital)
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No